CLINICAL TRIAL: NCT05062395
Title: Positron Emission Tomography for the Diagnosis of Immune Checkpoint Inhibitor-Related Myocarditis
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0206; NCI-2021-00838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0206 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-25; First posted 2021-09-30 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Myocarditis Acute
MeSH Terms: interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endomyocardial biopsy specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (diet, FDG PET CT): Patients receive a low carbohydrate and high fat diet for 48-72 hours. Patients receive FDG then undergo PET CT.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Other: Low Carbohydrate High Fat Diet; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG PET CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Undergo FDG PET CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Low Carbohydrate High Fat Diet — low carbohydrate and high fat diet for 48-72 hours
Procedure: Positron Emission Tomography — Undergo FDG PET CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This study evaluates positron emission tomography for the diagnosis of immune checkpoint inhibitor-related myocarditis. Immune checkpoint inhibitors have shown promising results in various malignancies however, several immune related adverse events have been described of which myocarditis carries the highest reported mortality. Diagnostic procedures, such as positron emission tomography, help find and diagnose myocarditis and provide functional or disease activity information as opposed to the largely structural/anatomic information.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To prospectively evaluate the sensitivity, specificity, positive predictive value, and negative predictive value of fludeoxyglucose F-18 (18 fluorodeoxyglucose) positive emission tomography computed tomography (PET CT) for the diagnosis of immune checkpoint inhibitor (ICI) related myocarditis.

SECONDARY OBJECTIVES:

I. To explore the clinical presentation and disease course of ICI-related myocarditis which include presenting symptoms (chest pain, dyspnea, fatigue), time from ICI initiation to symptom onset, hospitalization duration, time to peak troponin levels, and peak troponin levels.

II. To evaluate biomarkers, including peak troponin, peak no probnp, admission troponin level, and admission nt probnp level, and imaging modalities of ICI-related myocarditis which include sensitivity, specificity, positive predictive value, and negative predictive value of cardiac magnetic resonance imaging (MRI).

III. To determine the response to various treatments of ICI-related myocarditis which include time to resolution of symptoms, hospitalization duration, and peak troponin value stratified by treatment.

IV. To observe the long-term outcomes, including late decline in left ventricular ejection fraction (LVEF) to < 50%, and survival after ICI related myocarditis, and monitoring of ICI-related myocarditis.

V. To assess differences in PET CT imaging results between patients on steroid therapy versus not on steroid therapy for myocarditis.

OUTLINE:

Patients receive a low carbohydrate and high fat diet for 48-72 hours. Patients receive 18 fluorodeoxyglucose (FDG) then undergo PET CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age >= 18 years
* Patients must be able to understand and be willing to sign a written informed consent document. Surrogate decision-makers of patients will be allowed to consent patients for this study
* Patients must be receiving or have a history of receiving any ICI therapy in monotherapy or combination therapy
* Patients must have a suspicion of ICI-related myocarditis either by clinical presentation, biomarkers, or other diagnostic modalities

Exclusion Criteria:

* Pregnant or lactating patients will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with ICI and presenting to the University of Texas MD Anderson Cancer Center (MDACC) with suspected ICI-related myocarditis
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value | through study completion, an average of a year.
  Calculations of sensitivity, specificity, positive predictive value, and negative predictive value and their 90% exact confidence intervals will be performed for the evaluation of positron emission tomography computed tomography considering endomyocardial biopsy as the gold standard. Secondary analysis of these parameters will be used considering the Bonaca et al diagnoses of immune checkpoint inhibitor (ICI)-related myocarditis as a new gold standard. Receiver operating characteristic (ROC) curve and the AUC value (area under the ROC curve) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas L Palaskas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org